CLINICAL TRIAL: NCT04374175
Title: SERum-bank for PANcreatic Cancer
Acronym: SERPAN
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 20CH035; 2020-A00393-36 (Other: ANSM)
Record Dates: First submitted 2020-04-28; First posted 2020-05-05 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Adenocarcinoma
Keywords: Adenocarcinoma; Pancreatic cancer; Adiponectin; Blood sample
MeSH Terms: conditions — Adenocarcinoma; Pancreatic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adenocarcinoma group: Patients with Adenocarcinoma will be included. They will have blood sample at the inclusion visit and at 3 months, 6 months, 9 months and 12 months after.
  Interventions: Biological: Blood sample
- Control group: Patient with no adenocarcinoma will be included. They will have blood sample at the inclusion visit.
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — Blood sample will be performed

SUMMARY:
This study is about pancreatic cancer. If the diagnostic cancer is done at an early stage (<2cm), the chances of recovery are very good.

But the main problem is there is not any detections means for this cancer. Sadly, when there is a cancer diagnostic , it's already too late in the majority of cases, because the cancer is in an advanced case.

Today, there is no any effective means of detection... Blood markers can be a simple means of early detection

DETAILED DESCRIPTION:
The purpose of this study is to establish a sero-library in a case-control cohort to assess several potentially useful serum biomarkers, such as adiponectin in the early diagnosis of pancreatic cancer.

ELIGIBILITY:
ADENOCARCINOMA GROUP

Inclusion Criteria:

* Documented adenocarcinoma (cytology / anatomopathology), all stages, except if the tumor is immediately resectable and does not require preoperative cytological evidence. In this case, the inclusion and the first collection of the sero bank is done preoperatively. The diagnostic confirmation will therefore be made post-operatively at the risk of being excluded in the event of a different diagnosis.
* At the start of treatment (before surgery / 1st course of chemotherapy)
* Age ≥ 18 years
* Patient affiliated or entitled to a social security system

Exclusion Criteria:

* Patient refusal
* Acute renal failure
* Child-Pugh B or C cirrhosis
* Patient under guardianship or curators
* Other synchronous cancer or history of cancer <5 years
* Language barrier

CONTROL GROUP

Inclusion Criteria:

* Age ≥ 40 years
* Patient affiliated or entitled to a social security system
* Digestive endoscopy for any reason other than cancer or chronic inflammatory bowel disease

Exclusion Criteria:

* Patient refusal
* Acute renal failure
* Child-Pugh B or C cirrhosis
* Patient under guardianship or curators
* Other synchronous cancer or history of cancer <5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There are 2 groups: patients with adenocarcinoma (ADENOCARCINOMA GROUP) and without (CONTROL GROUP)
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Serum adiponectin concentration | Months : 0
  Measure by blood sample result Serum adiponectin concentration threshold for which the specificity will be 100% for the diagnosis of pancreatic cancer with a sensitivity of 80%.

SECONDARY OUTCOMES:
Serum CA19.9 concentration | Months : 0, 3, 6, 9, 12
  Measure by blood sample result Threshold for Comparison of diagnostic performance compared to serum adiponectin concentration
Tumor response and progression rates according to RECIST v1.1 | Month 12
  Tumor response and progression rates defined according to RECIST v1.1 criteria according to a serum threshold of the prognostic biomarker to be identified by logistic regression analyzes.
Progression-free survival | Months : 24
Overall survival | Months : 24
Serum adiponectin concentration | Months : 3, 6, 9, 12
  Measure by blood sample result Serum adiponectin concentration to correlate with cancer progression or not.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas WILLIET, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (2):
- France (2):
  - CHU Saint-Etienne, Saint-Etienne
  - Institut Cancérologique Lucien Newirth (ICLN), Saint-Priest-en-Jarez

IPD SHARING:
Plan to Share IPD: No